CLINICAL TRIAL: NCT01629017
Title: Longitudinal Evaluation of Recipients of Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Long Term Effects On Recipients of Hematopoietic Stem Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-4134
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Blood and Marrow Transplant (BMT)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project allows for the systematic collection and analysis of long-term follow-up clinical parameters in children who have received a stem cell transplant. The data collected will assist in determining appropriate intervention and treatment plans for patients enrolled on this study. In addition, future patients may benefit by having the ability to anticipate problems and develop methods of prevention or early intervention.

DETAILED DESCRIPTION:
Primary Objective: Implement long-term follow-up guidelines for children, adolescents and young adults who are survivors of HSCT while establishing a database which captures the survivor's lifetime care.

Secondary Objectives:

* Collect evidence-based data through a structured framework of periodic physical examination, laboratory and medical tests to monitor late effects in our HSCT survivors.
* Establish standards of care for late effects of therapy post HSCT for malignant and non-malignant diagnoses.
* Provide early identification and intervention towards recognized problems, as well as consistent education to foster a healthy lifestyle to all survivors.
* Collect blood and tissue samples to study immune reconstitution of all immune cell types and learn more about immune reconstitution and its affect on post-HSCT complications and disease free survival.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to receive OR has received a hematopoietic stem cell transplant (HSCT) for any condition.
* Participant may have had a HSCT in another institution than Lucile Packard Children's Hospital (LPCH) yet has transferred follow-up long-term care to our institution and is being seen through the late-effects clinic from the Pediatric HSCT program.
* Participant AND/OR parent/legally authorized representative is able to provide written informed consent and assent (as applicable) for participation.

Exclusion Criteria:

* Participant has relapsed from a malignant diagnosis post HSCT and is not being worked-up for a new HSCT.
* Participant or patient's authorized guardian is unable to provide consent and assent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Stanford Blood and Marrow Transplant clinic.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 1995-01; Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

PRIMARY OUTCOMES:
Collection of data and tissue samples with the goal of establishing a systematic follow-up care for HSCT recipients and a comprehensive database which can capture the particularities of survivors' clinical status through their life span. | This research study is expected to continue as long as we continue to perform clinical trials for children with diseases that involve the bone marrow or are affected by bone marrow production.

CONTACTS AND LOCATIONS:
Overall Officials: Ami Shah, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No